CLINICAL TRIAL: NCT03722654
Title: Measurement Training and Feedback System for Implementation of Family Therapy and CBT for Adolescent Externalizing Problems
Brief Title: Measurement Training and Feedback System: Family Therapy and CBT
Acronym: MTFS-FT-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH117212 (NIH)
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Adolescent Behavior
Keywords: Adolescents; Conduct problems; Delinquency; Substance misuse
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTFS (Experimental): MTFS-I Installation
  Interventions: Behavioral: MTFS-I Installation
- Control (No Intervention)

INTERVENTIONS:
Behavioral: MTFS-I Installation — MTFS-I Installation will focus on introducing MTFS-I components including weekly training modules and mock video segments to be coded, as well as monthly feedback reports summarizing therapist self-reported FT and CBT implementation in active cases. Facilitation will also be included to review progress and provide regular support.
  Arms: MTFS

SUMMARY:
This study aims to advance the science of mental health services for adolescent externalizing problems (AEPs) by developing therapist training procedures to increase fidelity to evidence-based interventions (EBIs) in usual care. Two widely endorsed approaches are consistently effective for treating AEPs: family therapy and CBT. Importantly, stronger fidelity to core EBIs of these approaches predicts better outcomes in research and community settings. Yet these EBIs are not widely implemented with fidelity. To help close this quality gap in adolescent services, investigators will develop an online intervention to strengthen fidelity to these EBIs in routine care: Measurement Training and Feedback System for implementation (MTFS-I). MTFS-I will target two essential aspects of EBI fidelity: Training components will seek to improve EBI self-monitoring, and a Feedback component will seek to increase EBI utilization. In keeping with NIMH's Experimental Therapeutics paradigm, this study will examine whether an Intervention (MTFS-I) has direct impact on immediate Targets (EBI self-monitoring and utilization).

If promising, future R01 studies will examine links among intervention, targets, and ultimate outcomes (AEPs). The MTFS-I package will be an online quality assurance system completed by therapists and supervisors that can be readily sustained in usual care. Two weekly Training components will adapt gold-standard observational fidelity coding procedures to promote improved self-monitoring of the targeted EBIs, and a monthly Feedback component will adapt a measurement feedback system to promote increased utilization of these EBIs in everyday practice. To maximize provider investment, sites will delineate their own fidelity standards for family therapy and CBT and help design feedback report templates.

The proposed study will be among the first to (1) test whether training therapists in observational assessment of EBI fidelity increases the accuracy with which they self-monitor use of those EBIs and (2) adapt measurement feedback procedures to track and improve therapist utilization of EBIs. To achieve study aims the investigators will first partner with two community clinics to develop sustainable MTFS-I procedures using a three-phase Pilot process. Investigators will then initiate an experimental Trial during which therapists (n = 32, treating 192 clients) at four different clinics will be randomized to MTFS-I versus no-intervention Control. In both conditions two kinds of data will be collected: therapist-report checklists on use of core family therapy and CBT techniques with adolescent cases and treatment session audio recordings. MTFS-I uptake will be tracked electronically for online components (Aim 1: MTFS feasibility). Session recordings will be coded by observers for three facets of EBI fidelity: adherence (extent of EBI utilization), working alliance, and therapist competence. Observer ratings will measure the strength of EBI self-monitoring (Aim 2: therapist reliability and accuracy) and fidelity (Aim 3 [EBI utilization] & Aim 4 [alliance, competence]). If effective, MTFS-I could be adapted to promote EBI fidelity for a variety of clinical populations and approaches.

DETAILED DESCRIPTION:
Discovering and disseminating effective methods to improve the quality of available treatment services for adolescent externalizing problems is an urgent public health priority. Despite the strong legislative and policy focus on quality of care evident in the CHIP Reauthorization Act of 2009 and the Affordable Care Act of 2010, comprehensive reports underscore the enduring "quality chasm" between behavioral treatments proven in controlled research versus those commonly practiced in usual care. The quality gap is highly evident for adolescent externalizing problems (AEPs), which encompass serious conduct problems, delinquency, and substance misuse. AEPs are the most common adolescent behavioral issues in specialty care, which follows from high prevalence rates: conduct disorder has a 9.5% lifetime prevalence rate, and 19% of adolescents report past-year illicit drug use with 7% meeting criteria for psychiatric disorder. Yet standard treatment quality for AEPs is considered mediocre to inadequate due to a host of factors headlined by the absence or modest quality of evidence-based services, insufficient provider training, and little quality monitoring.

Two behavioral treatment approaches are prime candidates for upgrading the quality of AEP treatment services. Both family therapy (FT) and cognitive-behavioral therapy (CBT) have excellent efficacy evidence for AEPs in both research and community settings. Each has strong support for treating serious conduct problems, delinquency, and substance use, and each has several manualized versions proven efficacious across the AEP range. Due to this extensive evidence base, there is incentive from clinical providers and payers to deliver these approaches in routine care: Both are now approved for treating AEPs by federal and private insurance plans and by regulatory agencies that govern licensed treatment providers. Notably, therapists report that both approaches are highly valued in everyday practice.

By consensus, the most efficient pathway toward improving the quality of mental health services is to increase the adoption and delivery of evidence-based interventions (EBIs) in usual care. However, there is a caveat: For EBIs to be effective in frontline settings, they must be delivered with sufficient fidelity to the principles and procedures of the approaches they represent. This remains a most difficult challenge for which innovative solutions are sorely needed. With regard to AEPs, controlled studies have shown that strong fidelity to the FT and CBT approaches predicts improved client outcomes in both efficacy and effectiveness studies. Yet, at this time, neither FT nor CBT are widely implemented with fidelity in community clinics that treat AEPs. To promote EBI fidelity as a core virtue of the behavioral care system, the study team published a theoretical model in which EBI implementation is recognized as an essential driver of positive client outcomes. This model includes structural characteristics of care that directly influence both implementation and outcomes, as well as outcomes considered relevant within the "quality of care" framework. The middle section depicts elements of implementation that have proven salient for effective EBI delivery, including technical factors (adherence to core treatment techniques, therapist competence) and relational factors (e.g., alliance), given that both are related to outcomes. According to this model and similar others, EBI implementation fidelity is a multidimensional construct with three primary facets: Adherence (extent to which signature EBI techniques are utilized), Competence (skillfulness and responsiveness of EBI delivery), and Alliance (working relationship between provider and client). In AEP research, fidelity-outcome studies consistently find that stronger EBI adherence and stronger alliance predict better client outcomes. Evidence for competence-outcome effects is less consistent, in large part because competence remains difficult to operationalize reliably. According to this framework, innovations aimed at improving service quality should directly target EBI fidelity; stronger EBI fidelity will then boost client outcome.

ELIGIBILITY:
Inclusion Criteria:

* Therapists treating adolescents aged 12-21 at partnering treatment sites

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in EBI Fidelity: ITT-ABP Therapist-Report | Conclusion of every session for 1 year
  Inventory of Therapy Techniques for Adolescent Behavior Problems is a 24-item, post-session, therapist-report fidelity tool that meets key criteria for pragmatic measures: relevance to stakeholders, low burden, broad applicability, strong psychometrics, and useful for data-driven decision-making (actionable). It requires 2-3 minutes to complete and was derived from validated observational fidelity tools for manualized treatments via a stakeholder-informed instrument adaptation process. The FT and CBT items each measure the adherence (i.e., thoroughness and frequency) with which each technique was used based on a 5-point Likert-type scale: 0 = Not at all, 1 = A little bit, 2 = Moderately, 3 = Considerably, 4 = Extensively.

SECONDARY OUTCOMES:
EBI Fidelity: ITT-ABP Observational Version | Through study completion, approximately 1 year
  The ITT-ABP observational version mirrors the therapist-report version, with the addition of two items. To capture Competence, we will use a single item (identical 5-point scoring scale): "Please rate the extent to which you were skillful and responsive in today's session". Competence is difficult to judge reliably even for trained coders. Nonetheless, we have had moderate success in coding Competence with a single item for both EBIs via the observational version of ITT-ABP: ICC = .55 for FT and .56 for CBT, 58. To capture Alliance, we will use the VTAS-R Short Form, a 5-item observational measure of therapeutic alliance, defined as the collaborative working relationship in therapy. The VTAS-R Short Form has likewise shown strong internal consistency, high correlations with the full-length VTAS-R, and predictive validity for retention and clinical outcomes for AEPs.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Hogue, PhD, Principal Investigator — The Center on Addiction
Locations (3):
- United States (3):
  - Roberto Clemente Center, New York, New York
  - The LGBT Community Center, New York, New York
  - Montefiore, New York, New York

REFERENCES:
- [Derived] Hogue A, Bobek M, MacLean A, Porter N, Jensen-Doss A, Henderson CE. Measurement training and feedback system for implementation of evidence-based treatment for adolescent externalizing problems: protocol for a randomized trial of pragmatic clinician training. Trials. 2019 Dec 10;20(1):700. doi: 10.1186/s13063-019-3783-8. PMID 31822294